CLINICAL TRIAL: NCT01860638
Title: A Double-Blind, Placebo-Controlled, Randomised, Phase II Study Evaluating the Efficacy and Safety of Addition of Continuous Multiple Line Bevacizumab Treatment to Lomustine in Second (2nd)-Line Followed by Standard of Care (SOC) in Third (3rd)-Line and Beyond Compared to Addition of Placebo, Following First Progression of Disease (PD1) in Patients With Glioblastoma (GBM) After First (1st)-Line Treatment With Radiotherapy, Temozolomide and Bevacizumab
Brief Title: A Comparison of Continuous Bevacizumab (Avastin) Treatment or Placebo in Addition to Lomustine Followed by Standard of Care After Disease Progression in Participants With Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO28347; 2012-003138-17 (EudraCT Number)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Lomustine; Radiotherapy; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- First-Line Bevacizumab followed by Bevacizumab + Lomustine/SOC (Experimental): Participants will receive first-line treatment with radiotherapy, temozolomide, and bevacizumab. All three treatments will be given concurrently for the first 6 weeks, followed by 6 cycles (28 days each) of temozolomide plus bevacizumab, followed by bevacizumab monotherapy until PD1 or unacceptable toxicity. At PD1, participants randomized to bevacizumab will receive bevacizumab plus lomustine until PD2. Following PD2, participants will continue with blinded bevacizumab with the addition of appropriate SOC. Following PD3, for subsequent treatment lines blinded bevacizumab may continue or open-label bevacizumab may be given at the discretion of the investigator and the participant.
  Interventions: Drug: Bevacizumab; Drug: Lomustine; Radiation: Radiotherapy; Drug: Temozolomide; Drug: SOC Agent
- First-Line Bevacizumab followed by Placebo + Lomustine/SOC (Placebo Comparator): Participants will receive first-line treatment with radiotherapy, temozolomide, and bevacizumab. All three treatments will be given concurrently for the first 6 weeks, followed by 6 cycles (28 days each) of temozolomide plus bevacizumab, followed by bevacizumab monotherapy until PD1 or unacceptable toxicity. At PD1, participants randomized to placebo will receive placebo plus lomustine until PD2. Following PD2, participants will continue with blinded placebo with the addition of appropriate SOC. Following PD3, for subsequent treatment lines blinded bevacizumab may continue or open-label bevacizumab may be given at the discretion of the investigator and the participant.
  Interventions: Drug: Bevacizumab; Drug: Lomustine; Drug: Placebo; Radiation: Radiotherapy; Drug: Temozolomide; Drug: SOC Agent

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 10 milligrams per kilogram (mg/kg) intravenous (IV) every 2 weeks (Q2W) throughout the study, with the exception of bevacizumab monotherapy prior to PD1, which will be given as 15 mg/kg IV every 3 weeks (Q3W).
  Other Names: Avastin
Drug: Lomustine — Lomustine will be administered at a dose of 90 milligrams per square meter (mg/m^2) orally (PO) every 6 weeks (Q6W), with a cap of 160 milligrams (mg) per dose. In the absence of hematologic toxicity following the first dose, the second and subsequent doses may be increased to 110 mg/m^2 PO Q6W, with a cap of 200 mg per dose.
Drug: Placebo — Placebo will be administered via IV infusion, in a formulation matched to bevacizumab, Q2W after randomization.
  Arms: First-Line Bevacizumab followed by Placebo + Lomustine/SOC
Radiation: Radiotherapy — Radiotherapy will be administered for a total dose of 60 Gray (Gy), administered in 2-Gy fractions, 5 days per week for 6 weeks during first-line treatment.
Drug: Temozolomide — Temozolomide will be administered orally (PO) as 75 mg/m^2 per day for the first 6 weeks of first-line treatment (concurrent treatment), followed by 6 cycles (28 days each) as follows: 150 mg/m^2 per day for the first 5 days of Cycle 1, then 200 mg/m^2 per day (if permitted by the participant's hematological and non-hematological toxicity profile) for the first 5 days of Cycles 2-6.
Drug: SOC Agent — The choice of SOC agent will be at the discretion of investigator. The SOC agent will be administered during third-line treatment and subsequent lines, as per standard practice.

SUMMARY:
This multicenter, double-blind, placebo-controlled, randomized study will evaluate the efficacy and safety of the addition of bevacizumab treatment to lomustine (in 2nd-line [2L] treatment) and SOC (in 3rd-line [3L] and subsequent lines of treatment) following first-line disease progression (PD1) in participants with newly diagnosed glioblastoma. All enrolled participants will receive 1L treatment with radiotherapy, temozolomide, and bevacizumab. At PD1, eligible participants will be randomized (1:1) to receive 2L treatment with either bevacizumab plus lomustine or placebo plus lomustine. After second-line disease progression (PD2), participants will receive 3L treatment and will continue blinded bevacizumab or placebo with the addition of an SOC agent. Following third-line disease progression (PD3), participants will receive subsequent lines of treatment and will either continue blinded bevacizumab or placebo (at the discretion of the investigator), or switch to open-label bevacizumab (at the choice of the participant).

ELIGIBILITY:
Inclusion Criteria at Enrollment (before PD1):

* Newly diagnosed, histologically confirmed glioblastoma not previously treated with chemotherapy or radiotherapy
* If female and not postmenopausal (less than [<] 12 months of amenorrhea) or surgically sterile, must agree to use a highly effective contraceptive method during the treatment period and for at least 6 months after the last dose of study drug
* Karnofsky performance status (KPS) greater than or equal to (>/=) 60
* Mandatory tissue collection during pre-study surgery or biopsy for confirmation of the diagnosis and pathology
* Craniotomy or intracranial biopsy site must be adequately healed. Study treatment should be initiated > 28 days following the last surgical procedure

Inclusion Criteria at Randomization (following PD1):

* Documented PD1 according to RANO criteria
* Eligibility for second-line treatment with lomustine and bevacizumab as investigational medicinal products
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Bevacizumab well tolerated and not interrupted for longer than 60 days during first-line treatment
* Tissue submission among participants for whom operation/re-operation is indicated before second-line treatment starts; operation/re-operation performed >/=28 days after last bevacizumab administration and second-line treatment initiated >/=28 days after surgical wound healed
* Randomization within 28 days after PD1 among participants for whom operation/re-operation is not necessary
* First administration of second-line treatment no later than 2 days from randomization

Exclusion Criteria at Enrollment (before PD1):

* Any prior chemotherapy for glioblastoma and low-grade astrocytomas
* Any prior radiotherapy to the brain or prior radiotherapy resulting in a potential overlap in the radiation field
* Prior or current anti-angiogenic treatment
* Treatment with any other investigational drug within 28 days or 2 investigational agent half-lives (whichever is longer) prior to first study treatment
* Inadequate hematological, renal, or liver function
* Inadequately controlled hypertension
* Prior history of gastrointestinal perforation or abscess
* Clinically significant cardiovascular disease
* History or evidence of central nervous system disease unrelated to cancer unless adequately treated with standard medical therapy
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding
* Serious non-healing wound, active ulcer, or untreated bone fracture
* Known hypersensitivity to any component of bevacizumab/placebo or any of the study drugs
* Active infection requiring IV antibiotics at start of study treatment
* Other malignancy within 5 years prior to study enrollment, except for carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ treated with curative intent
* Pregnant or lactating women
* Participation in any other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2013-08-19 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization at PD1 until death from any cause or end of study (overall approximately 35 months)

SECONDARY OUTCOMES:
Percentage of Participants Alive at 6, 12, and 18 Months from Randomization | At 6, 12, and 18 months after randomization/PD1 (overall up to approximately 35 months)
Progression-Free Survival (PFS) on 2L Treatment According to Modified Response Assessment in Neuro-Oncology (RANO) Criteria | From first administration of randomized treatment until PD2 or death from any cause (overall approximately 18 months)
PFS on 3L Treatment According to Modified RANO Criteria | From first administration of randomized treatment until PD3 or death from any cause (overall approximately 35 months)
Restricted PFS on 3L Treatment According to Modified RANO Criteria | From first administration of treatment after PD2 until PD3 or death from any cause (overall approximately 26 months)
Percentage of Participants with 2L Objective Response of Complete Response (CR) or Partial Response (PR) According to Modified RANO Criteria | From randomization/PD1 until PD2, death, subsequent anticancer therapy, operation/re-operation for glioblastoma, or 13 weeks after last administration of 2L-treatment, whichever occurs first (approximately 18 months overall)
Percentage of Participants with 3L Objective Response of CR or PR According to Modified RANO Criteria | From PD2 until PD3, death, subsequent anticancer therapy, operation/re-operation for glioblastoma, or 13 weeks after last administration of study treatment, whichever occurs first (approximately 26 months overall)
Percentage of Participants with 2L Disease Control as CR, PR, or Stable Disease According to Modified RANO Criteria | From randomization/PD1 until PD2, death, subsequent anticancer therapy, operation/re-operation for glioblastoma, or 13 weeks after last administration of 2L-treatment, whichever occurs first (approximately 18 months overall)
Percentage of Participants with 3L Disease Control as CR, PR, or SD According to Modified RANO Criteria | From PD2/start of 3L-treatment until PD3, death, subsequent anticancer therapy, operation/re-operation for glioblastoma, or 13 weeks after last administration of 3L-treatment, whichever occurs first (approximately 26 months overall)
Duration of 2L Objective Response Assessed According to Modified RANO Criteria | From first occurrence of CR/PR after randomization/PD1 until PD2, death from any cause, subsequent anticancer therapy, whichever occurs first (approximately 18 months overall)
Duration of 3L Objective Response According to Modified RANO Criteria | From first occurrence of CR/PR after PD2 until PD3, subsequent anticancer therapy, or death from any cause, whichever occurs first (approximately 26 months overall)
Percentage of Participants with Adverse Events (AEs) | From baseline up to 30 days after last dose (up to 41 months overall)
1L Treatment: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 (C30) Global Health Status/Global QoL Scale Score | Baseline;Week(Wk)3,5;end of Wk6;Maintenance:Day(D)1 (Visit[V]1), D15 (V2) Cycles(C)1-6 Q4W;Monotherapy:V1-V44 Q3W;Safety Follow-up(FU) (30 days after last 1L dose);PD FUs(8 Wk after Safety FU [PD FU1],then every 12 Wk until PD1) (up to 41 months overall)
2L and 3L Treatment: Change From 2L Baseline in EORTC QLQ C30 Global Health Status/Global QoL Scale Score | 2L Baseline (2L treatment V1); 2L treatment: V2-V41 (Q2W) until PD2; 3L treatment: V1-V61 (Q2W) until PD3; Safety FU (30 days after last 3L dose); PD FU1 (8 Wk after Safety FU); end of study (up to 41 months overall)
1L Treatment: Change From Baseline in EORTC QLQ Brain Cancer Module 20 (BN20) Multiple Item Score | Baseline; Wk 3, 5; end of Wk6; Maintenance: D1(V1), D15(V2) of C1-6 (Q4W); Monotherapy: V1-V44 (Q3W); Safety FU (30 days after last 1L dose); PD FUs (8 Wk after Safety FU [PD FU1], then every 12 Wk until PD1) (up to 41 months overall)
2L and 3L Treatment: Change From 2L Baseline in EORTC QLQ BN20 Multiple Item Score | 2L Baseline (2L treatment V1); 2L treatment: V2-V41 (Q2W) until PD2; 3L treatment: V1-V61 (Q2W) until PD3; Safety FU (30 days after last 3L dose); PD FU1 (8 Wk after Safety FU); end of study (up to 41 months overall)
Percentage of Participants with Mini Mental Status Examination (MMSE) Score <27 or >/=27 | Baseline and 2L Baseline
1L Treatment: Change From Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) z-score | Baseline; Maintenance: D1(V1) Cycles 1, 3, 5 (Q4W); Monotherapy: every 3rd visit starting from V1 to V43 (Q3W); Safety FU (30 days after last 1L dose); PD FUs (8 Wk after Safety FU [PD FU1], then every 12 Wk until PD1) (up to 41 months overall)
2L and 3L Treatment: Change From 2L Baseline in HVLT-R z-score | 2L Baseline; 2L treatment: every 6th visit starting from V7 to V43 (Q2W); 3L treatment: every 6th visit starting from V1 to V37, V49, V61 (Q2W); Safety FU (30 days after last 3L dose); PD FU1 (8 Wk after Safety FU); end of study (up to 41 months overall)
1L Treatment: Change From Baseline in Controlled Oral Word Association (COWA) z-score | Baseline; Maintenance: D1(V1) Cycles 1, 3, 5 (Q4W); Monotherapy: every 3rd visit starting from V1 to V43 (Q3W); Safety FU (30 days after last 1L dose); PD FUs (8 Wk after Safety FU [PD FU1], then every 12 Wk until PD1) (up to 41 months overall)
2L and 3L Treatment: Change From 2L Baseline in COWA z-score | 2L Baseline; 2L treatment: every 6th visit starting from V7 to V43 (Q2W); 3L treatment: every 6th visit starting from V1 to V37, V49, V61 (Q2W); Safety FU (30 days after last 3L dose); PD FU1 (8 Wk after Safety FU); end of study (up to 41 months overall)
1L Treatment: Change From Baseline in Trail-Making Test (TMT) Part A and B z-score | Baseline; Maintenance: D1(V1) Cycles 1, 3, 5 (Q4W); Monotherapy: every 3rd visit starting from V1 to V43 (Q3W); Safety FU (30 days after last 1L dose); PD FUs (8 Wk after Safety FU [PD FU1], then every 12 Wk until PD1) (up to 41 months overall)
2L and 3L Treatment: Change From 2L Baseline in TMT Part A and Part B z-score | 2L Baseline; 2L treatment: every 6th visit starting from V7 to V43 (Q2W); 3L treatment: every 6th visit starting from V1 to V37, V49, V61 (Q2W); Safety FU (30 days after last 3L dose); PD FU1 (8 Wk after Safety FU); end of study (up to 41 months overall)
Number of Participants with Hospitalizations According to Type of Hospitalizations | From Baseline up to death or study withdrawal/study end (up to 41 months overall)
Duration of Hospitalizations According to Type of Hospitalizations | From Baseline up to death or study withdrawal/study end (up to 41 months overall)
EuroQol Five-Dimension Questionnaire (EQ-5D) Score | From Baseline up to death or study withdrawal/study end (up to 41 months overall)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (64):
- Austria (6):
  - Medizinische Universität Graz; Universitätsklinik für Neurologie, Graz
  - Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck; Department fuer Neurologie, Innsbruck
  - Kepler Universitätsklinikum GmbH - Neuromed Campus; Innere Medizin mit Neuroonkologie, Linz
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
  - Kaiser-Franz-Josef-Spital; Neurologische Abteilung, Vienna
- MBAL Serdika EOOD, Sofia, Bulgaria
- Canada (2):
  - Tom Baker Cancer Centre; Dept of Medicine, Calgary, Alberta
  - McGill University; Montreal Neurological Institute; Oncology, Montreal, Quebec
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Tartu University Hospital; Clinic of Hematology and Oncology, Tartu, Estonia
- France (11):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Hopital Avicenne; Neurologie, Bobigny
  - Hopital Saint Andre; Département de Radiothérapie Et D'Oncologie Médicale, Bordeaux
  - Hopital neurologique Pierre Wertheimer - CHU Lyon; Neurologie, Bron
  - Hopital Cote De Nacre; Unite Neurologie Generale, Caen
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Hopital Roger Salengro; Service de Neurologie, Lille
  - Hopital de La Timone - CHU de Marseille; Service de neuro-oncologie - Hôpital Adultes - 12ème étage, Marseille
  - Hôpital Central; Departement de Neuro-Oncologie, Nancy
  - Hopital Pitié Salpétrière - CHU; Service de neurologie 2 - Mazarin, Paris
  - Hopital Purpan, Toulouse
- Greece (3):
  - Agioi Anargyroi Anticancer Hospital; Radiotherapeutic Clinic, Kifissia
  - Hygeia Hospital, Marousi
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Italy (5):
  - Ospedale Bellaria; U.O. Oncologia Medica, Bologna, Emilia-Romagna
  - IFO - Istituto Regina Elena; Oncologia Medica, Rome, Lazio
  - Fondazione IRCCS Istituto Neurologico C. Besta; Neuro-oncologia Sperimentale e Terapia Genica, Milan, Lombardy
  - Azienda Ospedaliera Le Molintte di Torino; Dipartimento Di Neurologia - Oncologia, Turin, Piedmont
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Seconda, Padua, Veneto
- Riga East Clinical University hospital, Clinic Gailezers, Dept of Neurosurgery, Riga, Latvia
- Portugal (3):
  - IPO de Coimbra; Servico de Oncologia Medica, Coimbra
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - Hospital de Sao Joao; Servico de Oncologia, Porto
- Romania (3):
  - Institutul Oncologic Prof. Dr. Al. Trestioreanu Bucuresti, Bucharest
  - Institut Oncologic Ion Chiricuta; Departament Radioterapie, Cluj-Napoca
  - Spital Clinic Judetean Mures; Oncologie, Târgu Mureş
- Spain (15):
  - Hospital Universitario Son Espases; Servicio de Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - IInstituto Oncologico de San Sebastian, Oncologikoa; Servicio de Oncologia, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital Universitario Infanta Cristina; Servicio de Oncologia, Badajoz
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga
  - Hospital Clinico Universitario de Salamanca; Servicio de Oncologia, Salamanca
- Sweden (3):
  - Universitetssjukhuset; Onkologkliniken, Linköping
  - Norrlands Universitetssjukhus; Cancer Centrum, Umeå
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Turkey (Türkiye) (4):
  - Adana City Hospital, Medical Oncology, Adana
  - Baskent Universitesi Tıp Fakultesi; Ic Hastalıkları Anabilim Dalı Tıbbi Onkoloji Bilim Dalı, Ankara
  - Dokuz Eylul Uni ; Medical Oncology, Izmir
  - Kocaeli University Faculty of Medicine; Medical oncology, İzmit
- United Kingdom (5):
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrookes Hospital; Dept of Oncology, Cambridge
  - University College Hospital; Department of Oncology, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Brandes AA, Gil-Gil M, Saran F, Carpentier AF, Nowak AK, Mason W, Zagonel V, Dubois F, Finocchiaro G, Fountzilas G, Cernea DM, Chinot O, Anghel R, Ghiringhelli F, Beauchesne P, Lombardi G, Franceschi E, Makrutzki M, Mpofu C, Urban HJ, Pichler J. A Randomized Phase II Trial (TAMIGA) Evaluating the Efficacy and Safety of Continuous Bevacizumab Through Multiple Lines of Treatment for Recurrent Glioblastoma. Oncologist. 2019 Apr;24(4):521-528. doi: 10.1634/theoncologist.2018-0290. Epub 2018 Sep 28. PMID 30266892
- [Derived] Brandes AA, Mason W, Pichler J, Nowak AK, Gil M, Saran F, Revil C, Lutiger B, Carpentier AF. Can bevacizumab prolong survival for glioblastoma patients through multiple lines of therapy? Future Oncol. 2014 May;10(7):1137-45. doi: 10.2217/fon.14.75. PMID 24947255